CLINICAL TRIAL: NCT02173561
Title: Group vs. Individual Cognitive Processing Therapy for Combat-related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); STRONG STAR Consortium (Unknown)
Responsible Party: Principal Investigator, Patricia Resick, Professor, Duke University
Organization: VA Boston Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0116-1
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Cognitive Processing Therapy; combat; military; CPT; group therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Cognitive Processing Therapy-Cognitive Only (Experimental)
  Interventions: Behavioral: Group Cognitive Processing Therapy-Cognitive Only
- Individual Cognitive Processing Therapy-Cognitive Only (Experimental)
  Interventions: Behavioral: Individual Cognitive Processing Therapy-Cognitive Only

INTERVENTIONS:
Behavioral: Group Cognitive Processing Therapy-Cognitive Only — Cognitive Processing Therapy-Cognitive Only version (CPT-C) is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT-C is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Sessions will be conducted in groups of 8-12 participants. Sessions will be conducted twice weekly for six weeks; each session is 90 minutes.
  Other Names: Group CPT-C
  Arms: Group Cognitive Processing Therapy-Cognitive Only
Behavioral: Individual Cognitive Processing Therapy-Cognitive Only — Cognitive Processing Therapy-Cognitive Only (CPT-C) is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Individual sessions will be conducted twice weekly for six weeks; each session is 60 minutes.
  Other Names: Individual CPT-C
  Arms: Individual Cognitive Processing Therapy-Cognitive Only

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to compare group and individual CPT-C for the treatment of PTSD in OIF/OEF military personnel.

DETAILED DESCRIPTION:
Estimates indicate that between 100,000 and 300,000 Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF) veterans are at significant risk for chronic post-traumatic stress disorder (PTSD), which can become a chronic disorder that impacts all areas of a person's life. PTSD treatment programs are being developed throughout the Department of Defense (DoD) and the Veterans Affairs (VA), but because of the large number of Service Members returning from deployment with PTSD, it is often necessary to provide psychotherapy in groups. Cognitive Processing Therapy (CPT), an evidence-based treatment for PTSD, was originally developed as a group-based intervention. However, group-based CPT treatment has never been systematically compared to individual CPT treatment. The public policy implications of the results of this trial are significant. If both treatment formats are equivalent or if group treatment is better, then group treatment would be a more efficient and cost-effective therapy modality in most cases. On the other hand, if individual therapy is found to be superior, the investment of greater resources into individual therapy will be justified in order to provide the most effective treatment for PTSD to military personnel. The purpose of this study is to compare group-administered CPT-Cognitive-only version (CPT-C) to individual CPT-C for the treatment of PTSD in OIF/OEF military personnel. Three hundred (300) adult male and female active-duty OIF/OEF military personnel over 18 years of age will be enrolled into this study. Participants will be randomized between group and individual CPT-C.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active duty, activated Reservist, or activated National Guard OIF/OEF military personnel or OIF/OEF veterans seeking treatment for PTSD
* Diagnosis of PTSD determined by a clinician-administered Posttraumatic Stress Scale (PSSI)
* Person has experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a military deployment in support of OIF/OEF. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.
* Be over the age of 18
* Speak and read English
* Be stable on any psychotropic medications they may be taking.

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention
* Active psychosis
* Moderate to severe brain damage (as determined by the inability to comprehend the baseline screening questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PTSD symptoms as measured by thePosttraumatic Stress Disorder Checklist-Stressor-specific Version (PCL-S) | Baseline, weekly during treatment, posttreatment, 6-month and 12-month follow-up
  PCL-S measures symptoms of posttraumatic stress disorder in response to a specific stressor.

SECONDARY OUTCOMES:
Change from baseline in depressive symptoms as measured by the Beck Depression Inventory-II | Baseline, weekly during treatment, posttreatment, 6-month, and 12-month follow-up
  The BDI-II is one of the most widely used instruments for measuring the severity of depressive symptoms. It consists of 21 items that assess both affective and somatic symptoms related to depression and depressive disorders. Each item is composed of four statements that reflect symptom severity. The statements are scaled from 0 (no disturbance) to 3 (maximal disturbance). Scores on all items are summed to obtain a total severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Resick, PhD, ABPP, Principal Investigator — Duke University
Locations (1):
- Fort Hood Army Base, Fort Hood, Texas, United States

REFERENCES:
- [Result] Resick PA, Wachen JS, Dondanville KA, Pruiksma KE, Yarvis JS, Peterson AL, Mintz J; and the STRONG STAR Consortium; Borah EV, Brundige A, Hembree EA, Litz BT, Roache JD, Young-McCaughan S. Effect of Group vs Individual Cognitive Processing Therapy in Active-Duty Military Seeking Treatment for Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):28-36. doi: 10.1001/jamapsychiatry.2016.2729. PMID 27893032
- [Derived] Pruiksma KE, Taylor DJ, Wachen JS, Straud CL, Hale WJ, Mintz J, Young-McCaughan S, Peterson AL, Yarvis JS, Borah EV, Dondanville KA, Litz BT, Resick PA. Self-reported sleep problems in active-duty US Army personnel receiving posttraumatic stress disorder treatment in group or individual formats: secondary analysis of a randomized clinical trial. J Clin Sleep Med. 2023 Aug 1;19(8):1389-1398. doi: 10.5664/jcsm.10584. PMID 36988304
- [Derived] Wachen JS, Mintz J, LoSavio ST, Kennedy JE, Hale WJ, Straud CL, Dondanville KA, Moring J, Blankenship AE, Vandiver R, Young-McCaughan S, Yarvis JS, Peterson AL, Resick PA; STRONG STAR Consortium. The impact of prior head injury on outcomes following group and individual cognitive processing therapy among military personnel. J Trauma Stress. 2022 Dec;35(6):1684-1695. doi: 10.1002/jts.22870. Epub 2022 Aug 29. PMID 36039506
- [Derived] Miles SR, Hale WJ, Mintz J, Wachen JS, Litz BT, Dondanville KA, Yarvis JS, Hembree EA, Young-McCaughan S, Peterson AL, Resick PA. Hyperarousal symptoms linger after successful PTSD treatment in active duty military. Psychol Trauma. 2023 Nov;15(8):1398-1405. doi: 10.1037/tra0001292. Epub 2022 Jul 28. PMID 35901423
- [Derived] Straud CL, Dondanville KA, Hale WJ, Wachen JS, Mintz J, Litz BT, Roache JD, Yarvis JS, Young-McCaughan S, Peterson AL, Resick PA; STRONG STAR Consortium. The Impact of Hazardous Drinking Among Active Duty Military With Posttraumatic Stress Disorder: Does Cognitive Processing Therapy Format Matter? J Trauma Stress. 2021 Feb;34(1):210-220. doi: 10.1002/jts.22609. Epub 2020 Oct 19. PMID 33078467
- See also: Related Info — http://www.strongstar.org